CLINICAL TRIAL: NCT00932321
Title: Open Label, Randomized, Comparator-Controlled Study of the Contraceptive Efficacy of Norethindrone Acetate (NA) and Ethinyl Estradiol (EE)
Brief Title: Study of Safety and Efficacy of an Oral Contraceptive
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Warner Chilcott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PR-03903
Record Dates: First submitted 2009-06-30; First posted 2009-07-03 (Estimated); Results first posted 2011-03-22 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Prevention of Pregnancy
Keywords: Contraception
MeSH Terms: interventions — Norethindrone Acetate; Ethinyl Estradiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 24 Day NA/EE (Experimental): Norethindrone acetate 1 mg /ethinyl estradiol 20 mcg for 24 days of each 28 day cycle
  Interventions: Drug: Norethindrone Acetate/Ethinyl Estradiol 24 Days
- 21 Day NA/EE (Active Comparator): Norethindrone acetate 1 mg/ethinyl estradiol 20 mcg for 21 days of each 28 day cycle
  Interventions: Drug: Norethindrone Acetate /Ethinyl Estradiol 21 Days

INTERVENTIONS:
Drug: Norethindrone Acetate/Ethinyl Estradiol 24 Days — One tablet per day for 24 days of each 28 day cycle followed by 4 placebo tablets
  Arms: 24 Day NA/EE
Drug: Norethindrone Acetate /Ethinyl Estradiol 21 Days — One tablet per day for 21 days of each 28 day cycle followed by 7 placebo tablets
  Other Names: 21 Day NA/EE
  Arms: 21 Day NA/EE

SUMMARY:
This is a comparative study. The primary objective of the study is to assess the efficacy of a low dose oral contraceptive in the prevention of pregnancy. The secondary objectives are to assess the incidence of intracyclic bleeding of norethindrone acetate/ethinyl estradiol (NETA/EE) administered for 24 days and NETA/EE administered for 21 days; and to assess the safety and tolerability of the product.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Women
* Age 18-45
* At risk for pregnancy
* History of regular cycles

Exclusion Criteria:

* Contraindications for use of hormonal contraception
* Conditions which affect the absorption or metabolism of steroid hormones
* BMI > 35

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 938 (Actual)
Dates: Start 2004-01; Primary Completion 2004-11 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herman Ellman, MD, Study Director — Sponsor GmbH
Locations (31):
- United States (31):
  - Warner Chilcott Investigational Site, Birmingham, Alabama
  - Warner Chilcott Investigational Site, Phoenix, Arizona
  - Warner Chilcott Investigational Site, Chico, California
  - Warner Chilcott Investigational Site, Los Angeles, California
  - Warner Chilcott Investigational Site, San Diego, California
  - Warner Chilcott Investigational Site, Denver, Colorado
  - Warner Chilcott Investigational Site, Boynton Beach, Florida
  - Warner Chilcott Investigational Site, Jacksonville, Florida
  - Warner Chilcott Investigational Site, Miami, Florida
  - Warner Chilcott Investigational Site, Palm Harbor, Florida
  - Warner Chilcott Investigational Site, Venice, Florida
  - Warner Chilcott Investigational Site, West Palm Beach, Florida
  - Warner Chilcott Investigational Site, Decatur, Georgia
  - Warner Chilcott Investigational Site, Powder Springs, Georgia
  - Warner Chilcott Investigational Site, Roswell, Georgia
  - Warner Chilcott Investigational Site, Savannah, Georgia
  - Warner Chilcott Investigational Site, Louisville, Kentucky
  - Warner Chilcott Investigational Site, Kansas City, Missouri
  - Warner Chilcott Investigational Site, St Louis, Missouri
  - Warner Chilcott Investigational Site, New Bern, North Carolina
  - Warner Chilcott Investigational Site, Winston-Salem, North Carolina
  - Warner Chilcott Investigational Site, Allentown, Pennsylvania
  - Warner Chilcott Investigational Site, Philadelphia, Pennsylvania
  - Warner Chilcott Investigational Site, Pittsburgh, Pennsylvania
  - Warner Chilcott Investigational Site, Charleston, South Carolina
  - Warner Chilcott Investigational Site, Greenville, South Carolina
  - Warner Chilcott Investigational Site, Sandy City, Utah
  - Warner Chilcott Investigational Site, Norfolk, Virginia
  - Warner Chilcott Investigational Site, Richmond, Virginia
  - Warner Chilcott Investigational Site, Virginia Beach, Virginia
  - Warner Chilcott Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 32 investigational study sites recruited 938 women aged 18 - 45 years of age beginning Feb '04
Pre-assignment Details: MITT Population defined as subset of All Treated Subjects who were evaluated for pregnancy, either positive or negative, at least once after beginning the study medication. Completed subjects - subset of MITT subjects completing at least 161 days of treatment based on returned drug or diary.
Groups:
- 24 Day NA/EE: Norethindrone acetate/ethinyl estradiol 1 tablet daily for 24 days followed by 4 placebo tablets
- 21 Day NA/EE: Norethindrone acetate/ethinyl estradiol 1 tablet daily for 21 days followed by 7 placebo tablets
Period: Overall Study
Arm/Group | 24 Day NA/EE | 21 Day NA/EE
Started | 751 | 187
MITT Population | 705 | 181
Completed | 580 | 141
Not Completed | 171 | 46

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24 Day NA/EE | 21 Day NA/EE | Total
Number analyzed (Participants) | 751 | 187 | 938
Age, Customized [Number; unit: Participants] — MITT (Modified Intent to Treat) Population
  Participants
    Age, Unknown | 1 | 1 | 2
    18-35 years | 579 | 151 | 730
    > 35 years | 125 | 29 | 154
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 751 | 187 | 938
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 751 | 187 | 938

OUTCOME MEASURES:

1. Primary Outcome: Pregnancy Rate (Expressed as Pearl Index) for Women 18 to 45 Years Old, MITT Population
Description: Pearl Index = 1300 * number of pregnancies/number of women-cycles of treatment
Time Frame: 5.6 months (6 - 28 day cycles)
Population: Modified intention to treat (MITT) subset of all treat subjects - evaluated for pregnancy at least once after beginning study medication.
Measure: Number; unit: Pearl Index
Arm/Group | 24 Day NA/EE | 21 Day NA/EE
Number analyzed (Participants) | 705 | 181
Pearl Index | 1.823 | 2.978

2. Secondary Outcome: Mean Number of Intracyclic Bleeding (IB)/Spotting Days in Cycles 2-6, MITT Population
Description: Self-reported via patient completed diary (none - no vaginal bleeding, light - less than normal menstruation, normal - like normal menstruation, heavy - more than normal menstruation) along with daily use of sanitary protection (other than panty liners). Light bleeding requiring no more than single pad or tampon will be spotting.
Time Frame: 5.6 months (6 - 28 day cycles)
Population: Modified Intent to Treat (MITT)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | 24 Day NA/EE | 21 Day NA/EE
Number analyzed (Participants) | 705 | 181
Days | 6.31 (9.16) | 7.31 (10.51)
Statistical Analysis 1: Comparison: 24 Day NA/EE vs 21 Day NA/EE; Test type: Non-Inferiority or Equivalence — Primary hypothesis tested was the independence (lack of association) of mean number of IB days in Cycles 2-6 across treatment groups; p = 0.311, Cochran-Mantel-Haenszel; Stratified by investigational site

ADVERSE EVENTS:
Time Frame: 10 months, between 5 Feb 2004 and 30 Nov 2004
Description: Nine randomized subjects returned all study medication unused resulting in the following treated subjects: 743 in 24 day NA/EE group and 186 in 21 day NA/EE group. Adverse Events were collected on this population.
Arm/Group | 24 Day NA/EE | 21 Day NA/EE
Serious Adverse Events (participants affected / at risk) | 3/743 | 0/186
Other Adverse Events (participants affected / at risk) | 457/743 | 99/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24 Day NA/EE (N=743) | 21 Day NA/EE (N=186)
Partial Thyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 24 Day NA/EE (N=743) | 21 Day NA/EE (N=186)
Headache (Nervous system disorders) | 47 | 13
Vaginal Candidiasis (Infections and infestations) | 45 | 10
Upper Respiratory Tract Infection (Infections and infestations) | 38 | 9
Sinusitis (Infections and infestations) | 23 | 4
Vaginitis bacterial (Infections and infestations) | 23 | 3
Urinary Tract Infection (Infections and infestations) | 18 | 5
Pharyngitis streptococcal (Infections and infestations) | 11 | 2
Gastroenteritis, Viral (Infections and infestations) | 8 | 4
Nausea (Gastrointestinal disorders) | 34 | 6
Vomiting (Gastrointestinal disorders) | 14 | 1
Diarrhea (Gastrointestinal disorders) | 9 | 1
Dyspepsia (Gastrointestinal disorders) | 8 | 2
Dysmenorrhea (Reproductive system and breast disorders) | 33 | 5
Breast Tenderness (Reproductive system and breast disorders) | 25 | 2
Metorrhagia (Reproductive system and breast disorders) | 14 | 2
Pelvic Pain (Reproductive system and breast disorders) | 10 | 2
Smear Cervix Abnormal (Investigations) | 23 | 6
Weight Increased (Investigations) | 15 | 3
Acne (Skin and subcutaneous tissue disorders) | 20 | 5
Mood Swings (Psychiatric disorders) | 16 | 5
Depression (Psychiatric disorders) | 8 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Fatigue (General disorders) | 8 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less